CLINICAL TRIAL: NCT04768309
Title: Assessment of the Production of Uremic Toxins by the Gut Microbiota of Patients With Chronic Kidney Disease: in Vitro Test
Brief Title: Impact of Intestinal Microbiota on Uremic Toxins Productions
Acronym: GUTCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_1078
Record Dates: First submitted 2021-02-12; First posted 2021-02-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: CKD; Uremia
Keywords: CKD; uremic toxin; probiotics; intestinal microbiota; artificial intestine
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD group (Experimental): CKD adult patients stage 4-5 Without diabetes BMI between 18 and 30 kg/m2
  Interventions: Other: Ex vivo exploration of the effect of a probiotic over precursor indole production
- Healthy volunteers group (Other): Adult without chronic treatment, without renal dysfunction
  Interventions: Other: Ex vivo exploration of the effect of a probiotic over precursor indole production

INTERVENTIONS:
Other: Ex vivo exploration of the effect of a probiotic over precursor indole production — Fresh feces in chronic kidney patients and healthy volunteers will be collected. The feces will be instilled in artificial intestine with and without selected probiotics and production of uremic toxins will be measured.

SUMMARY:
Chronic renal failure (CKD) affects 3 million people in France and is characterized by the accumulation of uremic toxins (UTs) such as p-cresyl sulfate (PCS) and indoxyl sulfate (IS) which participate in cardiovascular complications and disturbance of the carbohydrate metabolism associated with CKD. These UTs are not eliminated by dialysis due to their high affinity for albumin and alternative strategies to dialysis must be developed to decrease the production of TUs in patients not yet in dialysis. The dysregulation of the intestinal microbiota observed during CKD increases the generation of UTs in the intestine, by the transformation of amino acids derived from proteins (such as tyrosine and tryptophan transformed respectively into PCS and, IS). Thus, modulation of the intestinal microbiota seems to be an attractive target for reducing the production of UTs and the comorbidities associated with CKD. Some studies have demonstrated the potential interest of probiotics in lowering the plasma concentration of UTs, but the effects remain unclear. In order to test the interest of probiotics during CKD, the investigators have, in collaboration with the Nestlé laboratory and the ProDigest platform, the possibility of testing probiotics using a human intestine simulator before the investigation of experimental and human models. For this the investigators would need a collection of fresh stools. The fresh stools will be instilled in artificial intestine to test the efficacy of selected probiotics on UTs production.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Non diabetic (fasting blood glucose <1.26 g / L, or lack of insulin or oral antidiabetic treatment)
* BMI between 18 and 30 kg / m²
* Patient with CKD stage 4-5 ( eDFG < 30 ml/min/1.73m2 CKD-EPI)
* Not dialyzed
* No history of kidney transplant
* Patient followed in the nephrology department of Pr FOUQUE at the Lyon Sud hospital center

Exclusion Criteria:

* Active inflammatory, infectious, cardiovascular or neoplastic disease
* Colectomy, resection of the small intestine or cholecystectomy
* Patient having received antibiotics, prebiotics, probiotics in the last 3 months.
* Patient using laxatives (more than 2 doses per day for the last 3 months)
* Known renal pathology or known urologic malformation (healthy volunteer only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Production of precursor of one of major uremic toxins: indole | Indoles production will be measured 48 hours after instillation of fresh feces in the artificial intestine
  The main endpoint is the concentration of the precursor of indoxyl sulfate (indole) in the lumen of the artificial intestine with a microbiota of a patient with CKD compared to the concentration of indol in the lumen of artificial intestine with a microbiota from a patient with CKD and supplemented with a probiotic (supplied by Nestlé)

SECONDARY OUTCOMES:
Uremic toxins production | 48 hours after instillation of fresh feces in the human intestine simulator
  Concentration of various uremic toxins in a human intestine simulator (p-cresyl sulfate, p-cresol, indole-3-acetic acid, etc.).
Production of short-chain fatty acids (SCFA) | 48 hours after instillation of fresh feces in the human intestine simulator
  Concentration of short-chain fatty acids (SCFA) (acetate, propionate, butyrate, isobutyrate, isovalerate and isocaproate) human intestine simulator
Intestinal permeability in a human intestine simulator | 48 hours after instillation of fresh feces in the human intestine simulator
  It will be measured by the electrical transepithelial resistance of the intestinal cells.
Biochemical parameters | 48 hours after instillation of fresh feces in the human intestine simulator
  Concentration of ammonium and lactate in a human intestine simulator.
Biochemical parameters | 48 hours after instillation of fresh feces in the human intestine simulator
  pH levels of the human intestine simulator.
Biochemical parameters | 48 hours after instillation of fresh feces in the human intestine simulator
  Volume of gas production in a human intestine simulator.
Intestinal microbiota composition | 48 hours after instillation of fresh feces in the human intestine simulator
  Study of the composition of the intestinal microbiota by 16s analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Lyon Sud University Hospital, Pierre-Bénite, Rhône, France

REFERENCES:
- [Result] Beau A, Natividad J, Benoit B, Delerive P, Duboux S, Feng Y, Jammes M, Barnel C, Sequino G, Pinteur C, Glorieux G, Fouque D, Vidal H, Koppe L. A specifically designed multi-biotic reduces uremic toxin generation and improves kidney function. Gut Microbes. 2025 Dec;17(1):2531202. doi: 10.1080/19490976.2025.2531202. Epub 2025 Jul 12. PMID 40650408